CLINICAL TRIAL: NCT04599478
Title: Pharmacological and Behavioral Treatments to Treat Loss-of-Control Eating and Improve Weight Outcomes After Bariatric Surgery: Acute (Stage 1)
Brief Title: Pharmacological and Behavioral Treatment After Bariatric Surgery: Acute (Stage 1)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000029057; R01DK126637-01 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Loss-of-control Eating; Obesity/Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Naltrexone; bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Behavioral Weight Loss (BWL) + Naltrexone and Bupropion (NB) medication (Experimental): Participants randomly assigned to this arm will receive 16 weeks of BWL counseling and NB medication. The naltrexone and bupropion will be taken daily in pill form.
  Interventions: Drug: Naltrexone and Bupropion medication; Behavioral: Behavioral Weight Loss
- BWL + Placebo (Experimental): Participants randomly assigned to this arm will receive 16 weeks of BWL counseling and placebo. Placebo will be inactive and taken daily in pill form.
  Interventions: Behavioral: Behavioral Weight Loss; Other: Placebo
- NB medication (Experimental): Participants randomly assigned to this arm will receive 16 weeks of NB medication taken daily in pill form.
  Interventions: Drug: Naltrexone and Bupropion medication
- Placebo (Placebo Comparator): Participants randomly assigned to this arm will receive 16 weeks of placebo. Placebo will be inactive and taken daily in pill form.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naltrexone and Bupropion medication — NB medication will be taken daily in pill form.
  Other Names: Contrave
  Arms: Behavioral Weight Loss (BWL) + Naltrexone and Bupropion (NB) medication; NB medication
Behavioral: Behavioral Weight Loss — Behavioral Weight Loss (BWL) counseling includes weekly sessions.
  Arms: BWL + Placebo; Behavioral Weight Loss (BWL) + Naltrexone and Bupropion (NB) medication
Other: Placebo — Placebo will be inactive and taken daily in pill form.
  Arms: BWL + Placebo; Placebo

SUMMARY:
This study will compare the effectiveness of behavioral and pharmacologic treatments, alone and in combination, for the treatment of loss-of-control eating and weight following bariatric surgery. This is an acute treatment comparing behavioral weight loss alone or in combination with combination naltrexone/bupropion medication.

DETAILED DESCRIPTION:
Participants who provide informed consent and are determined to be eligible will then participate in the study.

A total of 160 patients with obesity and regular LOC-eating following MBS will be randomly assigned (double-blind) in a balanced factorial (2 X 2) design, to one of four 16-week interventions: BWL+NB, BWL+Placebo, NB, or Placebo. The randomization will be in equal proportions but stratified by surgery type.

ELIGIBILITY:
Inclusion Criteria:

* Be in the age range ≥18 years of age and ≤70 years of age.
* Have a BMI ≥30 (or BMI ≥27 with a medical comorbidity) and ≤50
* Have had laparoscopic Roux-en-Y gastric bypass or sleeve gastrectomy
* Approximately six months post-surgery
* Experience regular loss-of-control eating (defined as at least once weekly over the past 28 days)
* Be an otherwise healthy subject without uncontrolled medical problems, as determined by the study physician and medical co-investigators (physical examination, laboratory studies).
* Read, comprehend, and write English at a sufficient level to complete study-related materials.
* Provide a signed and dated written informed consent prior to study participation.

Be available for participation in the study for up to 19 months (7-month treatment plus 12-month follow up).

Exclusion Criteria:

* Has a predisposition to seizures (e.g., subject with a history or evidence of seizure disorder, febrile seizures during childhood, brain tumor, cerebrovascular disease, or significant head trauma; has a family history of idiopathic seizure disorder or is currently being treated with medications or treatment regimens that lower seizure threshold).
* Has a history of anorexia nervosa or history of bulimia nervosa.
* Is currently taking a medication that is a contraindication to NB medication (e.g., MAOI, opiates).
* Is currently using other medications for weight loss.
* Has a history of allergy or sensitivity to bupropion or naltrexone.
* Has a co-existing psychiatric condition that requires hospitalization or more intensive treatment (such as bipolar mood disorders, psychotic illnesses, or severe depression)
* Has untreated hypertension with a seated systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg, or heart rate > 100 beats/minute.
* Has a history of congenital heart disease, cardiovascular disease, cardiac arrhythmias requiring medication, or a history of cerebrovascular pathology including stroke.
* Has current uncontrolled hypertension.
* Has current uncontrolled Type I or Type II diabetes mellitus.
* Has untreated hypothyroidism with a TSH > 1.5 times the upper limit of normal for the test laboratory with repeat value that also exceeds this limit.
* Has gallbladder disease.
* Has a history of severe renal, hepatic, neurological, chronic pulmonary disease, or any other unstable medical disorder.
* Has a recent history of drug or alcohol dependence (since having bariatric surgery).
* Is currently in active treatment for eating or weight loss.
* Is currently participating in another clinical study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
* Is breast-feeding or is pregnant or is not using a reliable form of birth control.
* Reports active suicidal or homicidal ideation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Loss-of-control Eating Frequency | Post-treatment (4 months)
  Loss-of-control eating frequency is a continuous variable of loss-of-control eating episodes assessed using the Eating Disorder Examination interview; Loss-of-control eating frequency will be based on the past 28 days and defined as loss-of-control eating episodes per month.
Body Mass Index | Post-treatment (4 months)
  BMI is calculated using measured height and weight

SECONDARY OUTCOMES:
Loss-of-control Eating Remission | Post-treatment (4 months)
  Categorical: zero episodes/28 days
Weight loss | Post-treatment (4 months)
  Categorical: 5% weight loss
Eating Disorder Psychopathology | Post-treatment (4 months)
  Eating-disorder psychopathology is a continuous variable as assessed by the global score of the Eating Disorder Examination/Eating Disorder Examination-Questionnaire. Scores range from 0-6 (0=no eating-disorder psychopathology; 6=severe eating-disorder psychopathology).
Depressive Symptoms | Post-treatment (4 months)
  Depressive symptoms is a continuous variable of depressive symptomatology as assessed by the self-report measure, the Patient Health Questionnaire - 9. Scores range from 0-27 (0=no depressive symptoms, 27=greater depressive symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Department of Psychiatry, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No